CLINICAL TRIAL: NCT03295461
Title: Effect of Emblica Officinalis (Amla) as an Adjunct to Scaling and Root Planing in Patients With Chronic Periodontitis
Brief Title: Emblica Officinalis Irrigation in Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: perio shikha amla
Record Dates: First submitted 2017-09-25; First posted 2017-09-27 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- test group (Active Comparator): SRP+ 10% Emblica officinalis irrigation
  Interventions: Procedure: SRP+ 10% Emblica officinalis irrigation
- positive control group (Active Comparator): SRP + 0.2% Chlorhexidine irrigation
  Interventions: Procedure: SRP + 0.2% Chlorhexidine irrigation)
- negative control group (Active Comparator): SRP + 0.9% Saline irrigation
  Interventions: Procedure: SRP + 0.9% Saline irrigation
- test gropup (Active Comparator): SRP +10% E. officinalis gel application
  Interventions: Procedure: SRP +10% E. officinalis gel application.
- control group (Placebo Comparator): received SRP+ placebo gel application.
  Interventions: Procedure: SRP+ placebo gel application.

INTERVENTIONS:
Procedure: SRP+ 10% Emblica officinalis irrigation
  Arms: test group
Procedure: SRP + 0.2% Chlorhexidine irrigation)
  Arms: positive control group
Procedure: SRP + 0.9% Saline irrigation
  Arms: negative control group
Procedure: SRP +10% E. officinalis gel application.
  Arms: test gropup
Procedure: SRP+ placebo gel application.
  Arms: control group

SUMMARY:
E. officinalis fruit possesses both the antimicrobial and anti-inflammatory activities that may prove to be useful against several periodontal diseases with the advantage that it is devoid of side effects associated with synthetic drugs. After the careful search of literature, none of the studies have reported the effect of local drug delivery of E. officinalis preparations on chronic periodontitis.The present study is designed with the aim of assessing the effectiveness of Emblica officinalis extract formulations as a potential adjunctive therapeutic strategy in the management of chronic periodontititis

DETAILED DESCRIPTION:
The presence of bacterial plaque represents the principal etiologic factor involved in the initiation of inflammatory periodontal diseases and the destructive host responses triggered by microbial pathogens exaggerate the already existing condition resulting in connective tissue loss characterizing the inflammatory periodontal diseases . The key element of periodontal therapy is to achieve a significant reduction or eradication of suspected periodontal pathogens as well as modulation of destructive host responses.

Chlorhexidine has been extensively employed adjunctive to conventional mechanical treatment for chronic periodontitis. But its use is limited by various side effects, including development of resistance, decrease in saliva secretion, acceleration in calculus accumulation, altered taste perception and teeth staining Researchers are increasingly turning their attention to phyto-therapeutic agents and looking for new leads to develop better drugs against multidrug resistant microbial strains. Bacteria are less likely to develop resistance to these natural substances, which should be safer for patients and cause fewer side effects.

Emblica officinalis Gaertn. or Phyllanthus emblica Linn belongs to the family Euphorbiaceae. All parts of the plant are of use in treating various ailments, but the fruit is of immense use in various traditional systems of medicine as it possesses a wide array of activities such as antibacterial, anti-inflammatory, analgesic, antioxidant, immunomodulatory, antibacterial, antipyretic, antidiabetic, hypolipidaemic, cardioprotective, antiresorptive properties. E. officinalis fruit is one of the richest sources of Vitamin C (600mg/100g) and contains water, proteins, carbohydrates, fibres, minerals, zinc, chromium, copper, gallic acid. The antimicrobial property of E. officinalis fruit is attributed mainly to flavonoids, phenols, saponins and tannins. Saponins and tannins proved to have a potent anti-microbial property . Phenolic compounds of Emblica officinalis also ameliorate acute and chronic inflammation due to their modulatory action on free radicals and by affecting COX (Cyclo-oxygenase) pathway, specifically prostaglandins. Thus ,it was hypothesized that adjunctive use of E. officinalis along with nonsurgical periodontal treatment may improve periodontal tissue healing and /or treatment outcomes of chronic periodontitis.

Materials and methods:

The study was conducted in department of Periodontics and Oral Implantology, Post Graduate Institute of Dental Sciences (PGIDS), Rohtak in collaboration with College of Pharmacy and Department of Microbiology, Post Graduate Institute of Medical Sciences (PGIMS), Rohtak. This study was designed according to the ethical standards outlined in the 1964 Declaration of Helsinki, as revised in 2008. The study got approval from Institutional Review Board, PGIDS, Rohtak (PGIDS/2013/IEC/87) and ethical committee of PGIDS, Rohtak. The study continued from March 2013 to October 2014 and CONSORT guidelines for the randomized clinical trials were followed.

Study population: The study patients were enrolled from systemically healthy individuals attending regular outpatient department of Periodontics and Oral Implantology, PGIDS, Rohtak.

Study design included a single-center, double-blinded randomized clinical trial in two parts.

Part I :test group (n = 23, 264 sites) received scaling and root planing (SRP) +10% E.

officinalis gel application and control group (n = 23, 264 sites) received SRP+ placebo gel application.

Part II:test group (SRP+ 10% Emblica officinalis irrigation), positive control group (SRP + 0.2% Chlorhexidine irrigation), negative control group (SRP + 0.9% Saline irrigation)

Periodontal examination: After inclusion into the study, all patients underwent full-mouth periodontal examination in a standardized way using a mouth mirror, tweezer, Williams probe (Hu-Friedy, Chicago, IL.) and explorer. Following parameters were considered: Primary outcome variables including Probing Depth (PD), Clinical Attachment Level (CAL) and secondary outcome variables including Plaque Index (PI) , Gingival Index (GI) , Sulcus Bleeding Index (SBI) .

Preparation of E. officinalis extract: The authenticated plant material E.officinalis fruits (herbal garden, College of Pharmacy, Post Graduate Institute of Medical Sciences, Rohtak) were collected, washed and shade dried at room temperature. E. officinalis extract was prepared using the methodology according to Kokate, 2008 and 10% concentration of E. officinalis extract was finalized for subgingival gel/ irrigation in the present study.

Preparation of Emblica officinalis extract (Euphorbiaceae). The authenticated plant material E. officinalis fruits (herbal garden, College of Pharmacy, Post Graduate Institute of Medical Sciences, Rohtak) were collected, washed and shade dried at room temperature. A total of 500 g of powdered shade dried fruits of E. officinalis were extracted exhaustively with water and ethanol mixture without soaking. This suspension of powdered drug and hydroalcoholic mixture (1:1 ratio of water and ethanol) in sterile conical flask was then placed on magnetic stirrer at 50°C temperature for 4 h. Then the supernatant filtered by using Whatman filter paper, and the filterate was finely dried by using rotary film evaporator operating at 60 °C temperature and 75 rpm . This converted the extract into dried powder form, which was used for the gel formulation.

Preliminary antimicrobial and antiinflammatory screening - In this study, the authors assessed zones of inhibition and minimum inhibitory concentrations of E. officinalis hydroalcoholic extract against Streptococcus mutans (MTCC 497), Streptococcus oralis (MTCC 2696), Enterococcus fecalis (ATCC 29212), Pseudomonas aeruginosa (ATCC 27853) and Staphylococcus aureus (ATCC 25923) by agar diffusion and broth dilution tests, respectively. Zones of inhibition ranged between 10 and 28mm at 10% concentration of extract while minimum inhibitory concentration between 0.5% and 2% against tested micro-organisms. Antiinflammatory activity of extract was assessed by human red blood cell membrane stabilization method in vitro. Based upon these findings, 10%concentration of E. officinalis extract was finalized for subgingival application in the present study.

Periodontal treatment: Patients received non-surgical treatment in the form of full mouth supragingival and subgingival scaling and root planing (SRP) in 2-3 sessions .In part I of the study application of placebo gel and 10% E. officinalis gel in deep pockets of control and test group patients, respectively, in part II of the study singal application of subgingival irrigation with 0.9% saline, 0.2% chlorhexidine and 10% E. officinalis irrigant was performed in negative control group, positive control group and test group respectively, on the day of completion of SRP by another investigator (ST). The subgingival irrigation was accomplished by applying 5 ml irrigant to all the periodontal sites in both arches with the use of a syringe and blunted needle placed as close as possible to the bottom of the pocket. The patients were instructed to use only mechanical techniques to clean teeth during the study period and mouthwashes and /or antimicrobials were not prescribed. All the periodontal parameters were recorded at baseline and after 2 and 3 months of follow up period by a single periodontist (SG).

ELIGIBILITY:
Inclusion Criteria

:• systemically healthypatients with chronic periodontitis, at least eight sites with probing pocket depth (PPD) ≥5mm

* ≥30 years old,
* ≥ 20 teeth and .

Exclusion Criteria:

* presence of systemic illnesses (diabetes mellitus, immunocompromised states), which affect the outcome of periodontal therapy,
* history of periodontal therapy and use of antibiotics or antiinflammatory drugs in the preceding 6 months,
* allergy to gel components,
* aggressive periodontitis,
* pregnancy or lactation,
* smokers(current/former), alcohol or drug abuse.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
clinical attachment level | 3 MONTHS
  CAL

CONTACTS AND LOCATIONS:
Overall Officials: shikha Tewari, Study Director — POST GRADUATE INSTITUTE OF DENTAL SCIENCES
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No